CLINICAL TRIAL: NCT03472950
Title: Safety and Efficacy of Ranolazine for the Treatment of Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Jeffrey Statland, Assistant Professor, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00141491
Record Dates: First submitted 2018-03-01; First posted 2018-03-21 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: ALS
MeSH Terms: interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ranolazine 500mg (Experimental): Participants will take Ranolazine 500mg twice daily for up to 4 weeks.
  Interventions: Drug: Ranolazine 500 MG
- Ranolazine 1000mg (Experimental): Participants will take Ranolazine 1000mg twice daily for up to 4 weeks.
  Interventions: Drug: Ranolazine 1000 MG

INTERVENTIONS:
Drug: Ranolazine 500 MG — Ranolazine is an FDA approved drug for angina (ongoing chest pain or pressure that is felt when the heart does not get enough oxygen).
  Arms: Ranolazine 500mg
Drug: Ranolazine 1000 MG — Ranolazine is an FDA approved drug for angina (ongoing chest pain or pressure that is felt when the heart does not get enough oxygen).
  Arms: Ranolazine 1000mg

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of Ranolazine, and how well it is tolerated in patients with Amyotrophic Lateral Sclerosis (ALS). Ranolazine is an FDA approved drug that is used for decreasing chest pain.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a progressive debilitating and fatal neurodegenerative disease involving the motor neurons in the primary motor cortex, corticospinal tracts, brainstem and spinal cord with 5,000 newly diagnosed patients per year in the USA. There is a pressing need for additional therapies, as the only two FDA-approved drugs for ALS, riluzole and edaravone, showed prolongation of median survival of only two to three months and only a modest benefit in daily functioning, respectively. The ability to identify FDA approved drugs which can be repurposed to ALS, and which may slow disease progression, alleviate symptoms, or prolong survival will have an immediate positive impact of the lives of patients with ALS and their family members. Hypothesis: Ranolazine, an FDA approved drug for angina which inhibits the late Na+ current and intracellular Ca2+ accumulation may be neuroprotective in ALS by reducing neuronal hyperexcitability, may slow disease progression and reduce cramp frequency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically definite, probable, laboratory supported probable, or possible ALS per revised El Escorial criteria
* Cramp frequency greater than 4 cramps per week during 2 week run in
* ALS functional rating scale-revised (ALSFRS-R) score of greater than 24
* Able to lie on back for study procedures

Exclusion Criteria:

* Tracheostomy invasive ventilation, or use of non-invasive ventilation greater than 12 hours per day
* Pregnant or lactating
* Participation in a prior experimental drug trial less than 30 days prior to screening
* Patients taking ranolazine
* Patients taking medications which are contraindicated for use with ranolazine such as strong CYP3 inhibitors (ketoconazole, clarithromycin, nelfinavir), and CYP3 inducers (rifampin, phenobarbital)
* Patients with clinically significant medical comorbidities (hepatic, renal, cardiac, etc)
* Patients with baseline QT interval prolongation on Electrocardiography (ECG)
* Patients pre-disposed to secondary QT prolongation for other health conditions like family history of congenital long QT syndrome, heart failure, bradycardia, or cardiomyopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Statland, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg
Started | 6 | 8
Completed | 6 | 4
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 1 | 2 | 3
Age, Continuous [Median (Full Range); unit: years] | 53 [42 to 67] | 55 [39 to 71] | 54 [39 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 8 | 14
  Non Hispanic | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLT)
Description: Measured as any drug-related serious adverse event, or drug-related adverse event necessitating study withdrawal. If a dose has less than 33% DLTs it will be considered tolerable.
Time Frame: Up to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg
Number analyzed (Participants) | 6 | 8
Participants | 1 | 2

2. Secondary Outcome: Percent Change in Cramp Frequency
Description: The percent change in cramp frequency: average daily cramp frequency, comparing week 12-baseline
Time Frame: Weekly for 12 weeks
Measure: Mean (Standard Deviation); unit: Percent Change in Cramp Frequency
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg
Number analyzed (Participants) | 6 | 8
Percent Change in Cramp Frequency | -39.98 (23.94) | -68.38 (27.74)

3. Secondary Outcome: Percentage Change in Average Weekly Cramp Severity
Description: Percent change in average weekly cramp severity (1 being a very mild muscle cramp and 10 being the most severe cramp you ever experienced)
Time Frame: Weekly for 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change in average weekly cram
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg
Number analyzed (Participants) | 6 | 8
Percentage change in average weekly cram | -38.68 (19.46) | -54.05 (39.94)

4. Secondary Outcome: Change in Nocturnal Awakenings Per Week, Comparing Week 12 to Baseline
Time Frame: Weekly for 12 weeks
Measure: Mean (Standard Deviation); unit: Number of nights awakened
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg
Number analyzed (Participants) | 6 | 8
Number of nights awakened | -1.67 (2.09) | -4.57 (6.80)

5. Secondary Outcome: Muscle Fasciculations Count
Time Frame: Up to week 12
Measure: Mean (Standard Deviation); unit: Muscle fasciculations count
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg
Number analyzed (Participants) | 6 | 8
Muscle fasciculations count | 33 (25) | 58 (25)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 12 weeks. This began at baseline visit through the week 12 visit.
Arm/Group | Ranolazine 500mg | Ranolazine 1000mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine 500mg (N=6) | Ranolazine 1000mg (N=8)
Constipation (Gastrointestinal disorders) | 1 | 4
Gastroesophageal reflux (Gastrointestinal disorders) | 1 | 2
Dizziness (Ear and labyrinth disorders) | 0 | 1
Indigestion (Gastrointestinal disorders) | 0 | 1 (2)
Dental Abscess (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 0 | 2
Drowsiness (General disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Upper extremity weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Decreased muscle tone (Musculoskeletal and connective tissue disorders) | 0 | 1
Urine odor (Renal and urinary disorders) | 0 | 1
Worsening muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03472950/Prot_SAP_000.pdf